CLINICAL TRIAL: NCT06464744
Title: Investigating the Efficacy of rTMS Treatment in Improving Motor Function After Spinal Cord Injury: A Placebo-controlled Study
Brief Title: Efficacy of rTMS Treatment After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Mark Züchner, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 635283
Record Dates: First submitted 2024-06-05; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries; Myelopathy
Keywords: rTMS; rehabilitation; spinal cord injury; motor cortex stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Active motor cortex stimulation
Who Masked: Participant
Masking Description: Placebo motor cortex stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo stimulation (Placebo Comparator): Patients will receive stimulation from a placebo coil that only delivers skin tingling but no active brain stimulation.
  Interventions: Procedure: Placebo stimulation using a placebo coil
- Active stimulation (Active Comparator): Patients will receive active brain stimulation from a magnetic figure-of-eight-coil.
  Interventions: Procedure: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Procedure: Repetitive transcranial magnetic stimulation (rTMS) — Intermittent Theta burst stimulation will be delivered on the on the primary motor cortex using a figure-of-eight coil, supported by neuronavigation. The stimulation intensity will be set to 90% of the motor threshold
  Arms: Active stimulation
Procedure: Placebo stimulation using a placebo coil — The placebo coil looks identical to the active coil but it only delivers skin tingling and no active brain stimulation.
  Arms: Placebo stimulation

SUMMARY:
There is accumulating evidence that neuromodulation by repetitive transcranial magnetic stimulation (rTMS) of the motor cortex holds promise as a treatment for rehabilitation of motor function following a spinal cord injury. This study is designed to assess the clinical potential of non-invasive stimulation of the primary motor cortex to improve motor functions.The results will help to evaluate the clinical relevance of motor cortex stimulation for motor functions in patients with spinal cord injury. The outcomes of this study could potentially support the initiation of a larger clinical trial and the development of a new routine treatment.

DETAILED DESCRIPTION:
The investigators will recruit 20 patients with low cervical or thoracic ASIA C or D spinal cord injuries based on specific inclusion and exclusion criteria. The patients will be randomized into 2 groups. Each group will receive either the theta burst stimulation or the placebo stimulation. rTMS will be delivered using a figure-of-eight coil positioned on the patient's head, targeting the leg area of the primary motor cortex. After the motor threshold (MT) is determined patients will receive a unilateral 90% subthreshold theta burst stimulation for 3 minutes The protocol includes 15 stimulation sessions over a 3-week period. The 12-week follow up consist of a series of electrophysiological and functional tests to assess upper and lower limb function bilaterally. Secondary outcomes include pain using the NRS scale, and self-reported evaluation of autonomic functions before, during, and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years and less than 80 years
* Chronic patients with an incomplete cervical and/or thoracic spinal cord injury (traumatic and non-traumatic) affecting upper and/or lower extremities (i.e., C4-T12 and classified as ASIA C or D) (Figure 138).
* Capable and willing to provide informed consent and able to adhere to the treatment schedule
* Patients who can be followed for the whole duration of the study

6.3 Exclusion criteria

* Contraindication to rTMS:

  * past severe head trauma
  * history of epilepsy or ongoing epilepsy
  * active cerebral tumor
  * intracranial hypertension
  * implanted ferromagnetic devices such as cardiac pacemaker and neurostimulator and cochlear implants
  * pregnancy or lactation.
* Any clinically significant or unstable medical or psychiatric disorder
* Other ongoing research protocol or recent past protocol within two months before the inclusion
* History of treatment with Deep Brain Stimulation (DBS)
* Subjects protected by law (guardianship or tutelage measure)
* History of substance abuse (alcohol, drugs)
* Pending litigation
* Impossibility to understand the protocol or to fill out the forms
* Chronic use of sedative medication
* Participation in another clinical trial evaluating spinal cord injury

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Motor evoked potentials | From enrollment to the end of follow up at 12 weeks
  Motor evoked potentials will be recorded at the start and the end of each stimulation session.
Global spasticity | From enrollment to the end of follow-up at 12 weeks
  Spasticity will be evaluated by using the modified Ashworth scale from 0 (no spasticity) to 4 (rigid extremities).
Spasticity lower extremities | From enrollment to the end of follow-up at 12 weeks
  The Wartenberg pendulum is an objective test to assess the biomechanical properties of spasticity.The test consists of dropping the leg of a relaxed patient from a horizontal position and measuring oscillatory movements with a goniometer.
Nine-Hole Peg Test | From enrollment to the end of follow-up at 12 weeks
  The Nine-Hole Peg Test is used to measure manual dexterity in patients with various neurological diagnoses. It is described in the literature to explore upper extremity function. Patients are asked to take nine pegs (7 mm diameter, 32 mm length) from a container (square box measuring 100 x 100 x 10 mm), one by one, and place them into the holes on the board, as quickly as possible. Scores are based on the time taken to complete the test activity, recorded in seconds.
10-meter walking test | From enrollment to the end of follow-up at 12 weeks
  The 10-meter walk test (10MWT) is used to assess walking capabilities and walking speed in patients with gait impairments. Three trials will be recorded at the patient's fastest walking speed. The three trials are averaged and the gait speeds are documented in meters/second.
Lower extremities kinematics | From enrollment to the end of follow-up at 12 weeks
  Movement kinematics will be extracted from recordings with 3D motion capture trackers that will record joint coordinates in time.

SECONDARY OUTCOMES:
Numeric scale rating for pain evaluation | From enrollment to the end of follow-up at 12 weeks
  The analgesic efficacy of the stimulation protocol will be measured by the numeric scale rating (NRS), a self-reported measure in which patients rate their pain on a scale from 0 (no pain) to 10 (worst pain).
European myelopathy score | From enrollment to the end of follow-up at 12 weeks
  The European myelopathy score is a reliable tool to assess functional recovery. The score ranges from 5 to 18. Higher values indicate better neurological function (outcome).

OTHER OUTCOMES:
Potential adverse effect | From enrollment to the end of follow-up at 12 weeks
  In general, rTMS is a safe method. The use of exclusion criteria and ear plugs during stimulation will reduce side effects. Potential risks or side effects of rTMS include:
  * Displacement of ferromagnetic device
  * Headache (3% in conventional rTMS studies) because of the noise generated by the stimulation
  * Seizures (0,16% in conventional rTMS studies) particularly in those with past epilepsy or brain surgery
  * Application site pain or discomfort and jaw pain

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Atle Bjørnbeth, MD,PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital - Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No